CLINICAL TRIAL: NCT04593082
Title: Obesity as a Driver of Inflammation and Brain Volume Loss in Pediatric Multiple Sclerosis.
Brief Title: Obesity and Pediatric Multiple Sclerosis
Status: Recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, J. Nicholas Brenton, MD, Assistant Professor of Neurology and Pediatrics, University of Virginia
Other Study IDs: HSR200257
Record Dates: First submitted 2020-10-16; First posted 2020-10-19 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
Keywords: Pediatric; Obesity; Neurodegeneration; Inflammation
MeSH Terms: conditions — Multiple Sclerosis; Obesity; Nerve Degeneration; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric MS Subjects: Subjects with pediatric MS will undergo fasting lab work, non-contrasted MRI, DEXA scan, and surveys.
- Healthy controls: Non-MS pediatric control subjects who will undergo fasting lab work, DEXA scan, and surveys for comparison to control group.

SUMMARY:
Obesity is one possible contributor to severity of multiple sclerosis and progression of the disease. We already know that obesity is a risk determinant for acquiring MS, yet the impact of obesity on pediatric MS disease expression and course is unknown. This study will evaluate the relationship between obesity, obesity-derived inflammatory mediators, and imaging metrics of MS severity in children. Understanding how childhood obesity contributes to MS severity/progression may yield fundamental insights into disease pathobiology - which may thereby lead to effective strategies for halting its progression in its earliest stages.

ELIGIBILITY:
Pediatric MS subjects will meet below inclusion and exclusion criteria:

Inclusion Criteria:

* Ability to provide informed consent (or assent for minors)
* Relapsing-remitting MS diagnosis per 2017 McDonald criteria
* Ages ≥ 10 years to ≤ 20 years
* Diagnosis of MS or first clinical symptom of MS (whichever comes first) within ≤ 36 months from the time of enrollment.

Exclusion Criteria:

* Progressive form of MS
* Patients with an active, chronic disease of the immune system other than MS
* Conditions affecting the central nervous system (CNS) white matter (e.g. leukodystrophy) or for whom another condition may better explain imaging abnormalities (e.g. lupus)
* Myelin oligodendrocyte glycoprotein (MOG) antibodies on serologic testing
* Corticosteroid exposure within 30 days of study enrollment

Control subjects (Aim 2) will meet the below inclusion and exclusion criteria:

Inclusion Criteria:

* Ability to provide informed consent (or assent for minors)
* Age-, sex-, & BMI-matched to pediatric MS subjects (1:1 allocation)
* Healthy children and young adults from the local communities

Exclusion Criteria:

* History of past imaging or neurologic event raising concern for any inflammatory CNS process
* Medical history or previous/current diagnosis consistent with an autoimmune disorder pertaining to any system of the body (e.g. diabetes mellitus type 1, Crohn's disease, lupus)

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population will be draw from outpatient clinics at UVA and CHOP as well as the surrounding communities for each institution. Subjects will be screened for eligibility to include BMI measurements at time of study discussion if they are interested.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Whole brain volumes and focal demyelinating lesion volumes | 3 years
  58 patients with a recent MS diagnosis, stratified by weight category (29 normal weight and 29 overweight/obese). Subjects will undergo MRI to quantify total brain and lesion volume. Z-scores for volumetrics will be determined using age- and sex-matched normative data from the NIH-sponsored ABCD dataset. We will compare mean Z-scores of whole brain volume and focal demyelinating lesion volumes between the two groups.

SECONDARY OUTCOMES:
Adipo-cytokine profiles | 3 years
  Fasting adipo-cytokines from MS cohort will be compared to age-, sex-, and BMI-matched controls.
Adipo-cytokines correlation with brain volume loss and neuroaxonal injury | 3 years
  We will measure serum NfL in MS subjects and controls. We will determine if leptin (a pro-inflammatory adipo-cytokine) predicts degree of brain volume loss and/or neuroaxonal injury in subjects with MS. This exploratory, mechanistic aim has potential to provide the first link between obesity-derived inflammation and neuronal cell injury/loss.

CONTACTS AND LOCATIONS:
Overall Officials: J Nicholas Brenton, MD, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brenton JN, Koenig S, Goldman MD. Vitamin D status and age of onset of demyelinating disease. Mult Scler Relat Disord. 2014 Nov;3(6):684-8. doi: 10.1016/j.msard.2014.07.004. Epub 2014 Jul 28. PMID 25891547
- [Background] Woolbright EB, Brenton JN. Attitudes toward obestity and diet modification in pediatric MS patients. Americas Committee for Treatment and Research in Multiple Sclerosis (ACTRIMS); February, 28 2020, 2019; West Palm Beach, FL.
- [Background] Brenton JN, Woolbright E, Briscoe-Abath C, Qureshi A, Conaway M, Goldman MD. Body mass index trajectories in pediatric multiple sclerosis. Dev Med Child Neurol. 2019 Nov;61(11):1289-1294. doi: 10.1111/dmcn.14233. Epub 2019 Apr 5. PMID 30950520
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Centers for Disease Control. Healthy Weight. In. Vol 20162015
- [Background] Disanto G, Barro C, Benkert P, Naegelin Y, Schadelin S, Giardiello A, Zecca C, Blennow K, Zetterberg H, Leppert D, Kappos L, Gobbi C, Kuhle J; Swiss Multiple Sclerosis Cohort Study Group. Serum Neurofilament light: A biomarker of neuronal damage in multiple sclerosis. Ann Neurol. 2017 Jun;81(6):857-870. doi: 10.1002/ana.24954. PMID 28512753
- [Background] Chitnis T, Gonzalez C, Healy BC, Saxena S, Rosso M, Barro C, Michalak Z, Paul A, Kivisakk P, Diaz-Cruz C, Sattarnezhad N, Pierre IV, Glanz BI, Tomic D, Kropshofer H, Haring D, Leppert D, Kappos L, Bakshi R, Weiner HL, Kuhle J. Neurofilament light chain serum levels correlate with 10-year MRI outcomes in multiple sclerosis. Ann Clin Transl Neurol. 2018 Oct 16;5(12):1478-1491. doi: 10.1002/acn3.638. eCollection 2018 Dec. PMID 30564615
- [Background] Barro C, Benkert P, Disanto G, Tsagkas C, Amann M, Naegelin Y, Leppert D, Gobbi C, Granziera C, Yaldizli O, Michalak Z, Wuerfel J, Kappos L, Parmar K, Kuhle J. Serum neurofilament as a predictor of disease worsening and brain and spinal cord atrophy in multiple sclerosis. Brain. 2018 Aug 1;141(8):2382-2391. doi: 10.1093/brain/awy154. PMID 29860296
- [Background] Siller N, Kuhle J, Muthuraman M, Barro C, Uphaus T, Groppa S, Kappos L, Zipp F, Bittner S. Serum neurofilament light chain is a biomarker of acute and chronic neuronal damage in early multiple sclerosis. Mult Scler. 2019 Apr;25(5):678-686. doi: 10.1177/1352458518765666. Epub 2018 Mar 15. PMID 29542376
- [Background] Kuhle J, Nourbakhsh B, Grant D, Morant S, Barro C, Yaldizli O, Pelletier D, Giovannoni G, Waubant E, Gnanapavan S. Serum neurofilament is associated with progression of brain atrophy and disability in early MS. Neurology. 2017 Feb 28;88(9):826-831. doi: 10.1212/WNL.0000000000003653. Epub 2017 Feb 1. PMID 28148632
- [Background] Valcarcel AM, Linn KA, Vandekar SN, Satterthwaite TD, Muschelli J, Calabresi PA, Pham DL, Martin ML, Shinohara RT. MIMoSA: An Automated Method for Intermodal Segmentation Analysis of Multiple Sclerosis Brain Lesions. J Neuroimaging. 2018 Jul;28(4):389-398. doi: 10.1111/jon.12506. Epub 2018 Mar 8. PMID 29516669
- [Background] Shinohara RT, Sweeney EM, Goldsmith J, Shiee N, Mateen FJ, Calabresi PA, Jarso S, Pham DL, Reich DS, Crainiceanu CM; Australian Imaging Biomarkers Lifestyle Flagship Study of Ageing; Alzheimer's Disease Neuroimaging Initiative. Statistical normalization techniques for magnetic resonance imaging. Neuroimage Clin. 2014 Aug 15;6:9-19. doi: 10.1016/j.nicl.2014.08.008. eCollection 2014. PMID 25379412
- [Background] Hagler DJ Jr, Hatton S, Cornejo MD, Makowski C, Fair DA, Dick AS, Sutherland MT, Casey BJ, Barch DM, Harms MP, Watts R, Bjork JM, Garavan HP, Hilmer L, Pung CJ, Sicat CS, Kuperman J, Bartsch H, Xue F, Heitzeg MM, Laird AR, Trinh TT, Gonzalez R, Tapert SF, Riedel MC, Squeglia LM, Hyde LW, Rosenberg MD, Earl EA, Howlett KD, Baker FC, Soules M, Diaz J, de Leon OR, Thompson WK, Neale MC, Herting M, Sowell ER, Alvarez RP, Hawes SW, Sanchez M, Bodurka J, Breslin FJ, Morris AS, Paulus MP, Simmons WK, Polimeni JR, van der Kouwe A, Nencka AS, Gray KM, Pierpaoli C, Matochik JA, Noronha A, Aklin WM, Conway K, Glantz M, Hoffman E, Little R, Lopez M, Pariyadath V, Weiss SR, Wolff-Hughes DL, DelCarmen-Wiggins R, Feldstein Ewing SW, Miranda-Dominguez O, Nagel BJ, Perrone AJ, Sturgeon DT, Goldstone A, Pfefferbaum A, Pohl KM, Prouty D, Uban K, Bookheimer SY, Dapretto M, Galvan A, Bagot K, Giedd J, Infante MA, Jacobus J, Patrick K, Shilling PD, Desikan R, Li Y, Sugrue L, Banich MT, Friedman N, Hewitt JK, Hopfer C, Sakai J, Tanabe J, Cottler LB, Nixon SJ, Chang L, Cloak C, Ernst T, Reeves G, Kennedy DN, Heeringa S, Peltier S, Schulenberg J, Sripada C, Zucker RA, Iacono WG, Luciana M, Calabro FJ, Clark DB, Lewis DA, Luna B, Schirda C, Brima T, Foxe JJ, Freedman EG, Mruzek DW, Mason MJ, Huber R, McGlade E, Prescot A, Renshaw PF, Yurgelun-Todd DA, Allgaier NA, Dumas JA, Ivanova M, Potter A, Florsheim P, Larson C, Lisdahl K, Charness ME, Fuemmeler B, Hettema JM, Maes HH, Steinberg J, Anokhin AP, Glaser P, Heath AC, Madden PA, Baskin-Sommers A, Constable RT, Grant SJ, Dowling GJ, Brown SA, Jernigan TL, Dale AM. Image processing and analysis methods for the Adolescent Brain Cognitive Development Study. Neuroimage. 2019 Nov 15;202:116091. doi: 10.1016/j.neuroimage.2019.116091. Epub 2019 Aug 12. PMID 31415884
- [Background] Kerbrat A, Aubert-Broche B, Fonov V, Narayanan S, Sled JG, Arnold DA, Banwell B, Collins DL. Reduced head and brain size for age and disproportionately smaller thalami in child-onset MS. Neurology. 2012 Jan 17;78(3):194-201. doi: 10.1212/WNL.0b013e318240799a. Epub 2012 Jan 4. PMID 22218275
- [Background] Brenton JN, Koshiya H, Engel CE, Herrod S, Engelhard M, Goldman MD. Utility of Physical Disability Outcome Measures in Pediatric-Onset Multiples Sclerosis. American Academy of Neurology. 2017.
- [Background] Brenton JN, Koshiya H, Woolbright E, Goldman MD. The Multiple Sclerosis Functional Composite and Symbol Digit Modalities Test as outcome measures in pediatric multiple sclerosis. Mult Scler J Exp Transl Clin. 2019 Apr 29;5(2):2055217319846141. doi: 10.1177/2055217319846141. eCollection 2019 Apr-Jun. PMID 31065380
- [Background] Brenton JN, Woolbright E, Koshiya H, Engelhard M, Goldman MD. Continuous accelerometry as a measure of physical activity impairment in paediatric-onset multiple sclerosis subjects versus healthy controls. ECTRIMS Online Library. 2017
- [Background] Keyhanian K, Saxena S, Gombolay G, Healy BC, Misra M, Chitnis T. Adipokines are associated with pediatric multiple sclerosis risk and course. Mult Scler Relat Disord. 2019 Nov;36:101384. doi: 10.1016/j.msard.2019.101384. Epub 2019 Sep 5. PMID 31550559
- [Background] Castro K, Ntranos A, Amatruda M, Petracca M, Kosa P, Chen EY, Morstein J, Trauner D, Watson CT, Kiebish MA, Bielekova B, Inglese M, Katz Sand I, Casaccia P. Body Mass Index in Multiple Sclerosis modulates ceramide-induced DNA methylation and disease course. EBioMedicine. 2019 May;43:392-410. doi: 10.1016/j.ebiom.2019.03.087. Epub 2019 Apr 10. PMID 30981648
- [Background] Stampanoni Bassi M, Iezzi E, Buttari F, Gilio L, Simonelli I, Carbone F, Micillo T, De Rosa V, Sica F, Furlan R, Finardi A, Fantozzi R, Storto M, Bellantonio P, Pirollo P, Di Lemme S, Musella A, Mandolesi G, Centonze D, Matarese G. Obesity worsens central inflammation and disability in multiple sclerosis. Mult Scler. 2020 Sep;26(10):1237-1246. doi: 10.1177/1352458519853473. Epub 2019 Jun 4. PMID 31161863